CLINICAL TRIAL: NCT07089030
Title: A Pilot Study Evaluating the Benefit of Endoscopic Assessment for Iron Deficiency Anemia in Patients Receiving Antithrombotic Therapy
Brief Title: Endoscopic Evaluation for Iron Deficiency Anemia in Patients on Antithrombotic Therapy
Acronym: BEACON-IDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec (Other)
Responsible Party: Principal Investigator, Marie-Claude Lehoux, Principal Investigator, Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-708
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Obscure Gastrointestinal Bleeding; Iron-Deficiency Anemia; Antithrombotic Therapy
Keywords: Obscure Gastrointestinal Bleeding; Iron-Deficiency Anemia; Antithrombotic Therapy; Anticoagulants; Antiplatelet Agents; Endoscopy; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Anemia, Iron-Deficiency; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Endoscopic Evaluation (Active Comparator): Participants will undergo repeated gastrointestinal evaluations (e.g., endoscopy, colonoscopy, capsule endoscopy) as clinically indicated, along with iron supplementation (oral or IV) or blood transfusions as needed.
  Interventions: Procedure: Standard endoscopic evaluation
- Conservative Medical Management (Experimental): Participants will receive a single round of gastrointestinal evaluation, iron supplementation (oral or IV) or blood transfusions as needed, and regular lab monitoring (hemoglobin and ferritin levels).
  Interventions: Procedure: Conservative Medical Management

INTERVENTIONS:
Procedure: Standard endoscopic evaluation — Examinations of the gastrointestinal (GI) tract (including the stomach, small intestine, and colon) will be performed to identify the source of bleeding. These examinations may be repeated based on the treating physician's assessment. Iron supplementation (ferrous sulfate) will be administered either orally (per os) or intravenously (IV), and blood transfusions will be provided if necessary.
  Arms: Standard Endoscopic Evaluation
Procedure: Conservative Medical Management — The investigational intervention involves a conservative treatment approach guided by a decision-making algorithm based on iron deficiency anemia values. This algorithm, developed from guidelines by the British Society of Gastroenterology and the American Gastroenterological Association, determines whether patients receive oral or IV ferrous sulfate or a blood transfusion. Laboratory parameters (hemoglobin, ferritin) will be monitored at weeks 4, 12, 38, and 64. After iron therapy, hemoglobin response will be assessed at 4 weeks, and treatment will continue for ~3 months post-normalization to ensure iron store repletion. Blood tests will be repeated every 6 months to detect recurrence.
  Arms: Conservative Medical Management

SUMMARY:
This is a single-center, randomized pilot study evaluating the feasibility and safety of two management strategies for patients on antithrombotic therapy who present with obscure gastrointestinal bleeding (OGIB). Participants will be randomized to either repeated endoscopic evaluations or a conservative medical approach with limited testing. The study aims to assess whether conservative management yields similar clinical outcomes and quality of life compared to standard repeated endoscopic procedures. Results will inform the design of a larger trial and address the current lack of guidelines for managing recurrent iron-deficiency anemia in this patient population.

DETAILED DESCRIPTION:
Antithrombotic therapy plays a critical role in preventing thrombotic events in patients with atherosclerotic coronary artery disease and atrial fibrillation. However, these therapies are associated with an increased risk of gastrointestinal bleeding, including obscure gastrointestinal bleeding (OGIB), which is often recurrent and linked to high morbidity and mortality.

This single-center, prospective, randomized pilot study aims to assess the feasibility and safety of two different management strategies for patients on antithrombotic therapy presenting with OGIB. Approximately 20 participants will be randomized in a 1:1 ratio into two groups:

Group A will undergo repeated gastrointestinal evaluations (e.g., endoscopy, colonoscopy, capsule endoscopy) as clinically indicated, along with iron supplementation (oral or intravenous) or blood transfusions as needed.

Group B will receive a single round of gastrointestinal evaluation, iron supplementation or transfusions as needed, and regular laboratory monitoring (hemoglobin and ferritin levels).

The primary objective is to evaluate the feasibility of conducting a larger randomized controlled trial comparing conservative medical management to standard repeated endoscopic evaluation. The secondary objective is to compare the quality of life between the two groups.

This study will also assess recruitment strategies, measurement tools, and the safety of a "watchful waiting" approach. Ultimately, the findings will help determine whether endoscopic evaluation provides clinical benefit in patients with iron-deficiency anemia on antithrombotic therapy who have had negative initial endoscopic workups. Currently, there are no established guidelines for managing recurrent iron-deficiency anemia in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and postmenopausal women with iron deficiency anemia, and premenopausal women with iron deficiency anemia and a negative gynecological evaluation;

   a. Laboratory-confirmed iron deficiency anemia (hemoglobin < 120 g/L for women, < 130 g/L for men, and ferritin < 30 ng/L);
2. Patients receiving anticoagulant or antiplatelet therapy
3. Negative esophagogastroduodenoscopy (EGD), colonoscopy, and capsule endoscopy for gastrointestinal bleeding within six months prior to study enrollment
4. Willing and able to provide written informed consent
5. Able to read and understand French

Exclusion Criteria:

1. Ongoing overt gastrointestinal bleeding
2. Acute coronary syndrome, acute neurological event, sepsis, or respiratory failure within the past week
3. Pregnant women
4. Known gastrointestinal or hematological malignancy
5. Contraindications to capsule endoscopy
6. History of bariatric surgery, gastrectomy, or segmental resection of the small intestine
7. Inability to take oral iron
8. Other sources of blood loss (e.g., urinary, gynecological, hematoma, hemolysis)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Participant Enrollment | 64 weeks
  This will be evaluated by the :
  - Proportion of eligible participants who consent and receive the allocated intervention; - Proportion of treated participants who complete both laboratory tests and the quality-of-life questionnaire twice during the study period.
Hemoglobin level | At weeks 4, 12, 38, and 64 following enrollment
  Relative change of hemoglobin
Hematocrit level | At weeks 4, 12, 38, and 64 following enrollment
  Relative change of hematocrit
Ferritin | At weeks 4, 12, 38, and 64 following enrollment
  Relative change of ferritin
Reticulocyte count | At weeks 4, 12, 38, and 64 following enrollment
  Relative change of Reticulocyte count
Serum iron | At weeks 4, 12, 38, and 64 following enrollment
  Relative change of serum level
Transferrin saturation | At weeks 4, 12, 38, and 64 following enrollment
  Relative change of transferrin saturation
Total number of blood transfusions | At weeks 4, 12, 38, and 64 following enrollment
  The cumulative count of all blood transfusion events administered to a participant during the study period.
Total number of dose of ferrous sulfate administered | At weeks 4, 12, 38, and 64 following enrollment
  The cumulative count of individual doses of ferrous sulfate given to a participant during the study period
Adverse Events Reporting | Continuously monitored and recorded throughout the 12-month follow-up period
  Adverse events will be documented in the case report form (CRF). Events will be classified as serious or non-serious. A serious adverse event is defined as any event resulting in hospitalization, including death from any cause, cardiovascular events related to anemia, or the occurrence of active bleeding. The need to discontinue antithrombotic therapy due to persistent anemia will also be recorded.

SECONDARY OUTCOMES:
Endoscopic Investigations and Diagnoses in the Standard Care Group | Throughout the 12-month follow-up period
  For participants in the standard care group, all endoscopic procedures performed (e.g., upper endoscopy, colonoscopy, capsule endoscopy) and any resulting diagnoses will be recorded. This information will be used to characterize the diagnostic yield and clinical management in the standard intervention arm.
Quality of Life Assessment (GIQLI) | At baseline and at week 64 (end of study)
  Quality of life will be assessed using the Gastrointestinal Quality of Life Index (GIQLI), a validated 36-item questionnaire developed in Germany. It includes five subscales: gastrointestinal symptoms, emotional well-being, physical function, social function, and medical treatment. Each item is scored from 0 to 4, with a total score ranging from 0 to 144. Higher scores indicate better quality of life. The validated French version of the GIQLI (Slim et al., 1999) will be used in this study. Completion time is approximately 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Éva Mathieu, PhD, Study Director — Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec
Locations (1):
- Centre hospitalier affilié universitaire régional de Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No